CLINICAL TRIAL: NCT07281898
Title: Efficacy of Burst Stimulation-Guided Ablation Strategy in Improving Single-Procedure Outcomes for Paroxysmal Atrial Fibrillation: A Multicenter, Prospective, Randomized Controlled Study
Brief Title: Burst Stimulation for Paroxysmal Atrial Fibrillation
Acronym: Burst-PAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhibing Lu (Other)
Responsible Party: Sponsor-Investigator, Zhibing Lu, The chief of cardiology department, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025198
Record Dates: First submitted 2025-11-23; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI) + Burst Stimulation + Individualized Linear Ablation
  Interventions: Procedure: Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI); Procedure: Burst Stimulation
- Control group (Active Comparator): Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI)
  Interventions: Procedure: Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI)

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI) — Pulmonary Vein Isolation (PVI) + Superior Vena Cava Isolation (SVCI)
Procedure: Burst Stimulation — Burst Stimulation + Individualized Linear Ablation
  Arms: Test group

SUMMARY:
Atrial fibrillation (AF) is one of the most common cardiac arrhythmias worldwide, associated with high morbidity and mortality rates. Epidemiological studies in China show that the prevalence of AF in individuals aged ≥60 years ranges from 2% to 3%, with rates continuing to rise due to population aging. Paroxysmal atrial fibrillation (PAF), if inadequately controlled, tends to progress to persistent AF, significantly increasing the risk of stroke, heart failure, and death. Catheter ablation has become a first-line therapy for drug-refractory PAF, with pulmonary vein isolation (PVI) recognized as the cornerstone procedure. However, multiple prospective studies and meta-analyses indicate that long-term recurrence rates following PVI alone remain as high as 30%-50%. This observation has prompted researchers to investigate the roles of non-pulmonary vein triggers, atrial remodeling, and electrophysiological substrate in PAF recurrence. The superior vena cava (SVC) has been identified as a common non-pulmonary vein trigger, with empirical SVC isolation demonstrating additional clinical benefits in select studies. Furthermore, the presence of atrial electrical remodeling and reentry-dependent substrate suggests that trigger-focused ablation strategies alone may be insufficient to prevent recurrence in certain PAF patients. Burst pacing-induced atrial tachyarrhythmias, such as atrial flutter or fibrillation, provide a practical method for assessing atrial substrate. Retrospective studies indicate that additional linear ablation targeting procedure-induced atrial tachycardias, such as typical atrial flutter, can significantly reduce PAF recurrence rates. However, this strategy currently lacks high-quality evidence from prospective randomized controlled trials.

To date, no large-scale randomized controlled trial (RCT) has systematically validated the impact of programmed burst pacing combined with individualized linear ablation on outcomes in PAF patients, nor have standardized induction protocols or supplementary ablation pathways been established. This study addresses a critical need for optimized treatment strategies in the field of catheter ablation, with significant clinical implications and potential for widespread application.

Therefore, this prospective, multicenter, randomized controlled trial aims to systematically evaluate the efficacy and safety of this strategy in reducing post-ablation PAF recurrence, improving quality of life, and controlling AF burden. The study seeks to fill the current evidence gap and advance AF treatment from standardized protocols toward individualized precision intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 80 years old;
* Documented diagnosis of paroxysmal atrial fibrillation (self-terminating and lasting < 7 days);
* Patients scheduled for initial radiofrequency catheter ablation (RFCA) treatment;
* Able to sign the informed consent form and comply with a minimum of 12 months of follow-up.

Exclusion Criteria:

* Presence of organic heart disease (e.g., rheumatic heart disease, severe valvular stenosis or regurgitation, post-valve replacement, or dilated cardiomyopathy);
* Concomitant atrial tachyarrhythmia requiring radiofrequency ablation (including typical atrial flutter and atrial tachycardia);
* Prior history of catheter ablation for any atrial tachyarrhythmia (including atrial fibrillation, atrial flutter, or atrial tachycardia);
* Concomitant hyperthyroidism, active malignant tumor, or other serious illness with a life expectancy of <1 year;
* Contraindications to anticoagulation;
* Inability to discontinue antiarrhythmic drugs for reasons other than atrial fibrillation;
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1-, 3-, 6-, 12-month follow-up

SECONDARY OUTCOMES:
The incidence of major adverse cardiovascular events (MACE), bleeding events, and all-cause mortality | perioperative period and 1-, 3-, 6-, 12-month follow-up
Rate of arrhythmia induction | intra-procedural
Incidence of complications | perioperative period and 1-, 3-, 6-, 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy of participants, the individual participant data (IPD) from this study will not be shared.